CLINICAL TRIAL: NCT03917147
Title: Correlation Between Hysteroscopic Diagnosis of Endometrial Hyperplasia and Histopathological Examination: a Prospective Cohort Study
Brief Title: Correlation Between Hysteroscopic Diagnosis of Endometrial Hyperplasia and Histopathological Examination
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Pasquale De Franciscis, Associate Professor, University of Campania Luigi Vanvitelli
Other Study IDs: N.592
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Endometrial Hyperplasia; Endometrial Neoplasms
Keywords: Endometrial Hyperplasia; Office Hysteroscopy; Predictive values; Sensitivity
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endometrial Biopsy

GROUPS / COHORTS (4):
- AUB in Post-Menopause: Abnormal Uterine Bleeding (AUB) in Post-Menopause
  Interventions: Procedure: Office Hysteroscopy
- Endometrial Thickening in post-menopause: Ultrasonographic detection of Thickened Endometrium in post-menopause
  Interventions: Procedure: Office Hysteroscopy
- Endometrial Thickening in pre-menopause: Ultrasonographic detection of Thickened Endometrium in pre-menopause
  Interventions: Procedure: Office Hysteroscopy
- Pharmacological history of Tamoxifen-related therapy regimens: Patients who had been treated with Tamoxifen
  Interventions: Procedure: Office Hysteroscopy

INTERVENTIONS:
Procedure: Office Hysteroscopy — Patients underwent office hysteroscopy with a 5-mm continuous-flow hysteroscope and endometrial biopsies were taken using miniaturized instruments. Histopathological examination was conducted to confirm the diagnosis.

SUMMARY:
A prospective cohort study at a Tertiary University Hospital. From January to December 2018, we enrolled women with the following criteria: abnormal uterine bleeding in post-menopause, endometrial thickening in pre-or post-menopause; tamoxifen usage. Patients underwent office hysteroscopy with a 5-mm continuous-flow hysteroscope and endometrial biopsies were taken using miniaturized instruments. Senior operators had to foresee histopathological diagnosis using a questionnaire. Histopathological examination was conducted to confirm the diagnosis.

DETAILED DESCRIPTION:
Patient underwent the procedure after the menstrual phase (day 6 to 10) of a spontaneous menstrual cycle. All the procedures were performed by means of a continuous flow small-diameter hysteroscope with oval profile (maximum diameter 5 mm, minimum diameter 3.9 mm) (Bettocchi Office Hysteroscope size 5, Karl Storz GmbH & Co., Tuttlingen, Germany) fitted with a 30-degree telescope of 2.9 mm gauge, using the vaginoscopic approach, without tenaculum and speculum, and using saline solution as distending medium at 90-100 mmHg pressure generated by a pneumatic cuff and measured by means of a manometer; the biopsies were performed with the "punch" or "grasp" technique using a 5 Fr grasping forceps inserted through the operating channel of the hysteroscope. In case of small intrauterine pathologies, they were easily removed by means of a straight bipolar electrode active by an electrosurgical generator (Versapoint II; Gynecare, Ethicon) used to provide a 50W power for the mildest vapour cutting mode (VC3).

The hysteroscopic diagnosis of hyperplasia was based on one or more of the following findings: (1) focal or diffuse, papillary or polypoid, endometrial thickening, (2) Abnormal vascular patterns; (3) evidence of glandular cysts; (4) abnormal architecture features of glandular outlets (thickening, irregular gland density, dilatation). Although no consensus or RCTs showed agreement in describing objective criteria for EH, several trials agreed on the previous morphologic evaluation. [8].

The procedures were taken by three senior gynaecologists (P.D.F, L.C., N.C) whose expertise and skills were equivalent. After every procedure, surgeons were asked to propose a suggestive histological categorization of the clinical diagnosis by means of a questionnaire, in order to standardize the assessment. The questionnaire was made of a progressive number which identified the biopsy and a multiple-choice question. Operators were asked to choose one from the following answers: Benign (including atrophic endometrium, proliferative endometrium, endometrial polyp/s); Endometrial Hyperplasia (simple or complex hyperplasia); Atypical Hyperplasia/Carcinoma (including atypical endometrial hyperplasia and adenocarcinoma) Biopsied histological samples were sent for histopathological analysis. The histopathological examination of all the specimens was performed at the Pathology Unit of University of Campania "Luigi Vanvitelli". Three senior gynecopathologists (INS), with the same skills and expertise, were addressed to evaluate all the biopsies

ELIGIBILITY:
Inclusion Criteria:

* abnormal uterine bleeding in post-menopause
* ultrasonographic detection of endometrial thickening in pre-menopause
* ultrasonographic detection of endometrial thickening in post-menopause
* follow-up after Tamoxifen-based therapy regimens

Exclusion Criteria:

* severe urinary symptoms
* history of severe comorbidities (autoimmune disorders, chronic diseases and severe cardiac disease)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women included in this study are referred by gynaecologists of the general outpatient rooms of the institution's hospital
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity For Endometrial Hyperplasia | 12 months
Correlation between histopathological and cllinical diagnosis for Endometrial Hyperplasia | 12 months

SECONDARY OUTCOMES:
Negative Predictive value | 12 months
Positive Predictive value | 12 months
Likelihood ratio | 12 months
Positive and negative post test probability | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Woman, Child and General and Specialized Surgery, University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghoubara A, Sundar S, Ewies AAA. Predictors of malignancy in endometrial polyps: study of 421 women with postmenopausal bleeding. Climacteric. 2018 Feb;21(1):82-87. doi: 10.1080/13697137.2017.1410783. Epub 2017 Dec 8. PMID 29219004
- [Background] Trimble CL, Kauderer J, Zaino R, Silverberg S, Lim PC, Burke JJ 2nd, Alberts D, Curtin J. Concurrent endometrial carcinoma in women with a biopsy diagnosis of atypical endometrial hyperplasia: a Gynecologic Oncology Group study. Cancer. 2006 Feb 15;106(4):812-9. doi: 10.1002/cncr.21650. PMID 16400639
- [Background] Bourdel N, Chauvet P, Tognazza E, Pereira B, Botchorishvili R, Canis M. Sampling in Atypical Endometrial Hyperplasia: Which Method Results in the Lowest Underestimation of Endometrial Cancer? A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2016 Jul-Aug;23(5):692-701. doi: 10.1016/j.jmig.2016.03.017. Epub 2016 Apr 4. PMID 27058769
- [Derived] De Franciscis P, Riemma G, Schiattarella A, Cobellis L, Guadagno M, Vitale SG, Mosca L, Cianci A, Colacurci N. Concordance between the Hysteroscopic Diagnosis of Endometrial Hyperplasia and Histopathological Examination. Diagnostics (Basel). 2019 Oct 7;9(4):142. doi: 10.3390/diagnostics9040142. PMID 31591361